CLINICAL TRIAL: NCT00094276
Title: Improving Asthma Care for Minority Children in Head Start
Brief Title: Intervention for Improving Asthma Care for Minority Children in Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 168; R01HL073833-01 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Breathmobile intervention combined with a Facilitated Asthma Communication intervention (FACI)
  Interventions: Behavioral: Facilitated Asthma Communication Intervention (FACI); Behavioral: Breathmobile intervention
- 2 (Active Comparator): FACI intervention
  Interventions: Behavioral: Facilitated Asthma Communication Intervention (FACI)
- 3 (Active Comparator): Breathmobile intervention
  Interventions: Behavioral: Breathmobile intervention
- 4 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Facilitated Asthma Communication Intervention (FACI) — A caregiver/PCP communication intervention designed to facilitate communication between parents and PCPs about a child's asthma severity and recommended therapy.
  Arms: 1; 2
Behavioral: Breathmobile intervention — A community-based service that is specifically designed to deliver asthma screening and special consultation directly to families and children in high-risk neighborhoods.
  Arms: 1; 3

SUMMARY:
This study will evaluate two interventions that are designed to reduce asthma morbidity and improve asthma care of children in Head Start in urban Baltimore.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma-related morbidity and mortality are disproportionately high among low-income African American children. The effects of asthma are particularly harsh in very young children and their families, resulting in high rates of emergency department care, hospitalization, decreased quality of life, and the risk of fatal asthma. Research suggests that the contributing factors to this high morbidity include under-use of asthma primary preventive care, sub-optimal medical management, and inappropriate asthma management behaviors. Despite the importance of early and regular asthma preventive care for children, this goal has proved elusive. Head Start programs offer an ideal venue for accessing high-risk, low-income preschool children and improving asthma morbidity. The study will test the hypothesis that removing barriers to preventive asthma care and facilitating communication between parents and primary care providers (PCP) are necessary prerequisites to optimally influence caregiver's asthma management practices. The study will remove barriers by the use of Breathmobile, a community-based service that is specifically designed to deliver asthma screening and special consultation directly to families and children in high-risk neighborhoods. In addition, the study will evaluate a caregiver/PCP communication intervention designed to facilitate communication between parents and PCPs about a child's asthma severity and recommended therapy.

DESIGN NARRATIVE:

This two times two modified factorial study design will compare the following in their effectiveness in reducing asthma morbidity and improving asthma management: a Breathmobile intervention combined with a Facilitated Asthma Communication intervention (FACI); a FACI alone; the Breathmobile intervention alone; or a control group. A total of 360 Head Start students ages 2 to 6 with symptomatic doctor-diagnosed asthma will be recruited. The primary study outcome measure will be the number of symptom-free days over a period of 12 months. Secondary outcomes include health care utilization (i.e., emergency department visits, hospitalizations, and primary care visits), asthma medications, parent asthma-related quality of life, parent asthma management practices, and cost-effectiveness. The study will test the hypothesis that a FACI combined with the Breathmobile intervention will be the most effective in improving parent and PCP management of the child's asthma and in reducing asthma morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma or reactive airway disease (RAD) OR
* Experienced asthma symptoms within 1 month prior to study entry
* Treated for asthma in the emergency department within 6 months prior to study entry
* Asthma symptoms include day or nighttime wheezing, shortness of breath and cough, or use of rescue medicine (e.g., albuterol or ventolin)

Exclusion Criteria:

* Currently participating in another asthma education research study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 336 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Symptom-free days | Measured at baseline, 6 months and 12 months

SECONDARY OUTCOMES:
Health care utilization (i.e., emergency department visits, hospitalizations, and primary care visits) | Measured at baseline, 6 months and 12 months
Asthma medications | Measured at baseline, 6 months and 12 months
Parent asthma-related quality of life | Measured at baseline, 6 months and 12 months
Parent asthma management practices | Measured at baseline, 6 months and 12 months
Cost-effectiveness | Measured at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S. Rand, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States